CLINICAL TRIAL: NCT04838730
Title: Influence of Clearing Open-capsule Device on Refractive Predictability in Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-0719
Record Dates: First submitted 2021-03-10; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental): Hanita CleaRing device (CE approved; AMAR Certificate)
  Interventions: Device: Surgical procedure

INTERVENTIONS:
Device: Surgical procedure — Standard cataract extraction procedure will be performed under local anesthesia (at physician discretion) and CleaRing device will be implanted together with SeeLens AF IOL.

SUMMARY:
CleaRing is intended to reduce posterior capsular opacification in cataract patients. The device is intended to be implanted together with standard posterior chamber IOL during cataract surgery.

DETAILED DESCRIPTION:
Study Design:

This study is a prospective, single-group, single-center, open-label study. Each study subject will be implanted with a CleaRing device together with SeeLens AF IOL in a single eye.

Study population:

Men and women designated for cataract surgery that meet the inclusion/exclusion criteria and provide written informed consent will be enrolled in the study.

Enrollment:

A total of 20 subjects will be enrolled.

Investigational sites:

Single-center study.

Duration of Subject participation:

The primary endpoint will be achieved when the study subject has completed a 1-month follow-up after the implantation of the CleaRing device.

Study Group:

Each subject will be implanted with a CleaRing device together with SeeLens AF IOL in a single eye.

Visits & Procedures Pre-operative visit: 0-3 months prior to the implantation procedure. The visit will include the subject's qualification assessment for inclusion/exclusion criteria as described above. Informed consent must be signed.

Complete anamnesis will be taken including the subject's medical complaints, medical history, medication use, and ophthalmic examinations.

Surgical procedure: Standard cataract extraction procedure will be performed under local anesthesia (at physician discretion) and CleaRing device will be implanted together with SeeLens AF IOL.

Follow-up: All subjects will have regular follow-up visits at the following post-operative periods: 1 day, 7 days, and 1 month. All postoperative visits will include a complete ophthalmic examination, a record of medications used, and documentation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

The subject is between 50 and 80 years of age The subject is designated for cataract surgery

Eye designated for the study fulfills the following criteria:

* Potentially able to achieve a good vision (by the opinion of the investigator)
* ACD is at least 2.5mm (from epithelium)
* Corneal astigmatism is at most 2.0 DPT
* Axial length is between 22.0 and 26.0 mm
* Able to obtain pupil dilation of at least 6.0 mm
* Average keratometry values between 42.0 and 46.0 D Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

1. Subject diagnosed with glaucoma of any type or having intraocular pressure above 24mmHg
2. Subject who has undergone previous intraocular surgery in eye designated for the study
3. Subject with a corneal abnormality that would prevent stable and reliable refraction
4. Subject with weak or torn zonules
5. Subject with Pseudoexfoliation syndrome (PEX)
6. Subject with amblyopia
7. Subject with a retinal disease that in the opinion of the principal investigator would prevent stable and reliable refraction or might be worsened due to implantation of the device
8. Subject is diagnosed with active anterior segment intraocular inflammation
9. Subject is obligated to previous participation in another study with any investigational drug or device within the past 30 days
10. Subject is pregnant

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
VISUAL ACUITY | 1 month
  Distance (far) manifest refraction and the testing distance used will be recorded on the case report forms. Manifest refraction will be determined using the maximum plus for best visual acuity method. The distance manifest refraction will be done with a distance adjusted chart but not less than 4 meters. The actual manifest refraction distance will be noted on the case report forms.
  Visual acuity will be measured with either Snellen or ETDRS format charts for distance.
  Results will be recorded in a LogMar scale.
SLIT LAMP EXAM | 1 month
  The slit lamp exam will include the measurement of aqueous cell and flare, and the measurement of corneal edema by a standard grading system. It will also include an evaluation for the presence of pupillary irregularities, iris atrophy and pigment dispersion, degree of posterior capsular opacification and correct position of the IOL and the CleaRing device.
  For the evaluation of aqueous cells and flare, use a slit lamp beam 0.3 mm wide and 1 mm high, and use the following grading:
  Cells none (0) = no cells seen trace (+1) = 1-5 cells seen mild (+2) = 6-15 cells seen moderate (+3) = 16-30 cells seen severe (+4) = > 30 cells seen
  Flare none (0) = No Tyndall effect trace (+1) = Tyndall effect barely discernible mild (+2) = Tyndall beam in anterior chamber is mildly intense moderate (+3) = Tyndall beam in anterior chamber is moderately intense severe (+4) = Tyndall beam is severely intense. The aqueous has a white and milky appearance.
MEASUREMENT OF INTRAOCULAR PRESSURE | 1 month
  Intraocular pressure will be measured using Goldmann applanation tonometry or other validated methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson, Holon, Israel